CLINICAL TRIAL: NCT03521934
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Effects of Sotagliflozin on Clinical Outcomes in Hemodynamically Stable Patients With Type 2 Diabetes POST Worsening Heart Failure
Brief Title: Effect of Sotagliflozin on Cardiovascular Events in Participants With Type 2 Diabetes Post Worsening Heart Failure (SOLOIST-WHF Trial)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to business decision
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15156; 2017-003510-16 (EudraCT Number); U1111-1190-7891 (Other: UTN)
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Results first posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotagliflozin (Experimental): Sotagliflozin 200 mg tablet once daily, with possible up-titration in the first 8 months to 400 mg, for up to 21.2 months.
  Interventions: Drug: Sotagliflozin
- Placebo (Placebo Comparator): Matching placebo to sotagliflozin 200 mg once daily, with possible up-titration in the first 8 months to matching placebo to sotagliflozin 400 mg, for up to 21.6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin — Pharmaceutical form: tablet
  Route of administration: oral
  Other Names: SAR439954
  Arms: Sotagliflozin
Drug: Placebo — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objective:

To compare the effect of sotagliflozin to placebo on the total occurrences of cardiovascular (CV) death, hospitalization for heart failure (HHF), and urgent visit for heart failure (HF) in hemodynamically stable participants after admission for worsening heart failure (WHF)

Secondary Objectives:

To compare the effects of sotagliflozin to placebo on:

* The total occurrences of HHF and urgent visit for HF
* The occurrence of CV death
* The occurrence of all-cause mortality
* The total occurrences of CV death, HHF, urgent visit for HF, non-fatal myocardial infarction (MI), and non-fatal stroke
* Change in Kansas City Cardiomyopathy Questionnaire-12(KCCQ-12) score
* Change in estimated glomerular filtration rate (eGFR)

DETAILED DESCRIPTION:
The estimated study duration for a given participants will be approximately 3 to 24 months.

ELIGIBILITY:
Inclusion criteria:

* Type 2 Diabetes Mellitus.
* Admitted to the hospital, or urgent heart failure visit for worsening heart failure.
* Prior diagnosis of heart failure (> 3 months).
* Prior chronic treatment for heart failure with a loop diuretic (eg furosemide, torsemide, bumetanide) for > 30 days.
* Randomized when hemodynamically stable, prior to hospital discharge or within 3 days of discharge.
* Brain natriuretic peptide (BNP) ≥150 picograms per milliliter (pg/mL) (≥450 pg/mL for participants with atrial fibrillation) or N-terminal B-type natriuretic peptide ≥600 pg/mL (≥1800 pg/mL for participants with atrial fibrillation).
* Participants with Left Ventricular Ejection Fraction <40% should be on beta-blockers and renin-angiotensin-aldosterone system (RAAS) inhibitors as per local guidelines unless contraindicated.
* Signed written informed consent.

Exclusion criteria:

* Age < 18 years or > 85 years.
* Worsening heart failure attributed to other causes such as pulmonary embolism, stroke, heart attack.
* Cardiac surgery or coronary procedure within 1 month or planned during study.
* Lower extremity complications (such as skin ulcer, infection, osteomyelitis, and gangrene) identified during screening and requiring treatment at randomization.
* Planning to start a sodium-glucose linked transporter-2 (SGLT2) inhibitor during the study.
* Acute coronary syndromes within 3 months prior to Randomization.
* Hemodynamically significant uncorrected primary valvular disease.
* Significant pulmonary disease contributing substantially to the participant's dyspnea.
* End stage Heart Failure.
* History of diabetic ketoacidosis (DKA) or nonketotic hyperosmolar coma within 3 months prior to screening.
* History of stroke within 3 months prior to randomization.
* History of dialysis within 1 year prior to randomization.
* History of solid organ transplant or on a transplant list (if heart transplant, defined as status 1 transplant).
* Severe kidney disease as defined by glomerular filtration rate (eGFR) <30 milliliter per minute per 1.72 meter square (mL/min/1.73 m^2).
* Pregnancy.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1222 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (466):
- United States (94):
  - Investigational Site Number 8400128, Alexander City, Alabama
  - Investigational Site Number 8400109, Cottonwood, Arizona
  - Investigational Site Number 8400032, Little Rock, Arkansas
  - Investigational Site Number 8400080, Little Rock, Arkansas
  - Investigational Site Number 8400075, Bakersfield, California
  - Investigational Site Number 8400069, Fresno, California
  - Investigational Site Number 8400008, Los Angeles, California
  - Investigational Site Number 8400063, Los Angeles, California
  - Investigational Site Number 8400127, National City, California
  - Investigational Site Number 8400007, Redondo Beach, California
  - Investigational Site Number 8400036, Stockton, California
  - Investigational Site Number 8400033, Sylmar, California
  - Investigational Site Number 8400049, Torrance, California
  - Investigational Site Number 8400028, Walnut Creek, California
  - Investigational Site Number 8400029, Bridgeport, Connecticut
  - Investigational Site Number 8400037, New Haven, Connecticut
  - Investigational Site Number 8400046, DeLand, Florida
  - Investigational Site Number 8400009, Gainesville, Florida
  - Investigational Site Number 8400079, Homestead, Florida
  - Investigational Site Number 8400031, Jacksonville, Florida
  - Investigational Site Number 8400022, Jacksonville, Florida
  - Investigational Site Number 8400098, Lake Mary, Florida
  - Investigational Site Number 8400058, Miami Beach, Florida
  - Investigational Site Number 8400105, Orlando, Florida
  - Investigational Site Number 8400082, Pensacola, Florida
  - Investigational Site Number 8400057, Port Charlotte, Florida
  - Investigational Site Number 8400006, Sarasota, Florida
  - Investigational Site Number 8400035, Tampa, Florida
  - Investigational Site Number 8400042, Tampa, Florida
  - Investigational Site Number 8400004, Wellington, Florida
  - Investigational Site Number 8400073, Atlanta, Georgia
  - Investigational Site Number 8400118, Tucker, Georgia
  - Investigational Site Number 8400067, Arlington Heights, Illinois
  - Investigational Site Number 8400043, Chicago, Illinois
  - Investigational Site Number 8400072, Elk Grove Village, Illinois
  - Investigational Site Number 8400055, Indianapolis, Indiana
  - Investigational Site Number 8400020, Muncie, Indiana
  - Investigational Site Number 8400122, Richmond, Indiana
  - Investigational Site Number 8400091, Waterloo, Iowa
  - Investigational Site Number 8400030, Covington, Louisiana
  - Investigational Site Number 8400065, Annapolis, Maryland
  - Investigational Site Number 8400012, Boston, Massachusetts
  - Investigational Site Number 8400001, Cambridge, Massachusetts
  - Investigational Site Number 8400077, Detroit, Michigan
  - Investigational Site Number 8400062, Kalamazoo, Michigan
  - Investigational Site Number 8400017, Kalamazoo, Michigan
  - Investigational Site Number 8400107, Duluth, Minnesota
  - Investigational Site Number 8400056, Jackson, Mississippi
  - Investigational Site Number 8400019, Columbia, Missouri
  - Investigational Site Number 8400103, Lee's Summit, Missouri
  - Investigational Site Number 8400132, Grand Island, Nebraska
  - Investigational Site Number 8400130, Lincoln, Nebraska
  - Investigational Site Number 8400083, Omaha, Nebraska
  - Investigational Site Number 8400071, Omaha, Nebraska
  - Investigational Site Number 8400015, Ridgewood, New Jersey
  - Investigational Site Number 8400050, Voorhees Township, New Jersey
  - Investigational Site Number 8400131, Albuquerque, New Mexico
  - Investigational Site Number 8400051, Brooklyn, New York
  - Investigational Site Number 8400111, Buffalo, New York
  - Investigational Site Number 8400097, The Bronx, New York
  - Investigational Site Number 8400061, The Bronx, New York
  - Investigational Site Number 8400045, Greensboro, North Carolina
  - Investigational Site Number 8400085, Raleigh, North Carolina
  - Investigational Site Number 8400078, Winston-Salem, North Carolina
  - Investigational Site Number 8400087, Cincinnati, Ohio
  - Investigational Site Number 8400047, Cincinnati, Ohio
  - Investigational Site Number 8400095, Maumee, Ohio
  - Investigational Site Number 8400099, Toledo, Ohio
  - Investigational Site Number 8400121, Zanesville, Ohio
  - Investigational Site Number 8400054, Arlington, Oregon
  - Investigational Site Number 8400134, Doylestown, Pennsylvania
  - Investigational Site Number 8400044, Natrona Heights, Pennsylvania
  - Investigational Site Number 8400115, Philadelphia, Pennsylvania
  - Investigational Site Number 8400039, Sayre, Pennsylvania
  - Investigational Site Number 8400114, Providence, Rhode Island
  - Investigational Site Number 8400100, Warwick, Rhode Island
  - Investigational Site Number 8400059, Charleston, South Carolina
  - Investigational Site Number 8400092, Columbia, South Carolina
  - Investigational Site Number 8400104, Greenville, South Carolina
  - Investigational Site Number 8400040, Rapid City, South Dakota
  - Investigational Site Number 8400088, Greenville, Tennessee
  - Investigational Site Number 8400089, Memphis, Tennessee
  - Investigational Site Number 8400053, Nashville, Tennessee
  - Investigational Site Number 8400041, Brownsville, Texas
  - Investigational Site Number 8400074, Dallas, Texas
  - Investigational Site Number 8400016, Houston, Texas
  - Investigational Site Number 8400123, McKinney, Texas
  - Investigational Site Number 8400101, New Braunfels, Texas
  - Investigational Site Number 8400066, Victoria, Texas
  - Investigational Site Number 8400093, Manassas, Virginia
  - Investigational Site Number 8400003, Richmond, Virginia
  - Investigational Site Number 8400126, Clarksburg, West Virginia
  - Investigational Site Number 8400038, Morgantown, West Virginia
  - Investigational Site Number 8400048, Manitowoc, Wisconsin
- Argentina (28):
  - Investigational Site Number 0320031, Caba
  - Investigational Site Number 0320009, Caba
  - Investigational Site Number 0320016, Capital Federal
  - Investigational Site Number 0320002, Ciudad de Buenos Aires
  - Investigational Site Number 0320022, Corrientes
  - Investigational Site Number 0320001, Corrientes
  - Investigational Site Number 0320024, Córdoba
  - Investigational Site Number 0320011, Córdoba
  - Investigational Site Number 0320003, Córdoba
  - Investigational Site Number 0320010, Córdoba
  - Investigational Site Number 0320025, Córdoba
  - Investigational Site Number 0320029, La Plata
  - Investigational Site Number 0320007, La Plata
  - Investigational Site Number 0320006, Merlo
  - Investigational Site Number 0320005, Morón
  - Investigational Site Number 0320012, Olivos
  - Investigational Site Number 0320023, Quilmes
  - Investigational Site Number 0320018, Rosario
  - Investigational Site Number 0320013, Rosario
  - Investigational Site Number 0320008, Salta
  - Investigational Site Number 0320020, San Martín
  - Investigational Site Number 0320028, San Miguel de Tucumán
  - Investigational Site Number 0320030, San Miguel de Tucumán
  - Investigational Site Number 0320019, San Miguel de Tucumán
  - Investigational Site Number 0320017, Santa Fe
  - Investigational Site Number 0320015, Santa Fe
  - Investigational Site Number 0320004, Villa Belgrano
  - Investigational Site Number 0320014, Villa María
- Australia (2):
  - Investigational Site Number 0360007, Murdoch
  - Investigational Site Number 0360001, Wollongong
- Austria (7):
  - Investigational Site Number 0400006, Braunau am Inn
  - Investigational Site Number 0400002, Feldkirch
  - Investigational Site Number 0400007, Graz
  - Investigational Site Number 0400005, Linz
  - Investigational Site Number 0400004, Salzburg
  - Investigational Site Number 0400003, Vienna
  - Investigational Site Number 0400001, Vienna
- Belgium (8):
  - Investigational Site Number 0560002, Aalst
  - Investigational Site Number 0560007, Ghent
  - Investigational Site Number 0560004, Kortrijk
  - Investigational Site Number 0560001, Leuven
  - Investigational Site Number 0560003, Liège
  - Investigational Site Number 0560005, Mol
  - Investigational Site Number 0560006, Mons
  - Investigational Site Number 0560008, Roeselare
- Brazil (19):
  - Investigational Site Number 0760009, Belo Horizonte
  - Investigational Site Number 0760024, Belo Horizonte
  - Investigational Site Number 0760002, Blumenau
  - Investigational Site Number 0760011, Brasília
  - Investigational Site Number 0760005, Campinas
  - Investigational Site Number 0760006, Campinas
  - Investigational Site Number 0760023, Fortaleza
  - Investigational Site Number 0760018, Goiânia
  - Investigational Site Number 0760010, Passo Fundo
  - Investigational Site Number 0760003, Porto Alegre
  - Investigational Site Number 0760020, Porto Alegre
  - Investigational Site Number 0760021, Porto Alegre
  - Investigational Site Number 0760007, Porto Alegre
  - Investigational Site Number 0760013, Porto Alegre
  - Investigational Site Number 0760004, Recife
  - Investigational Site Number 0760001, São José do Rio Preto
  - Investigational Site Number 0760012, São Paulo
  - Investigational Site Number 0760008, São Paulo
  - Investigational Site Number 0760017, Votuporanga
- Canada (13):
  - Investigational Site Number 1240013, Cambridge
  - Investigational Site Number 1240006, Granby
  - Investigational Site Number 1240015, Halifax
  - Investigational Site Number 1240002, Montreal
  - Investigational Site Number 1240019, Montreal
  - Investigational Site Number 1240018, Montreal
  - Investigational Site Number 1240004, Peterborough
  - Investigational Site Number 1240014, Québec
  - Investigational Site Number 1240007, Scarborough
  - Investigational Site Number 1240005, Sherbrooke
  - Investigational Site Number 1240011, Toronto
  - Investigational Site Number 1240001, Toronto
  - Investigational Site Number 1240009, Trois-Rivières
- Chile (11):
  - Investigational Site Number 1520009, Concepción
  - Investigational Site Number 1520011, Santiago
  - Investigational Site Number 1520006, Santiago
  - Investigational Site Number 1520003, Santiago
  - Investigational Site Number 1520004, Santiago
  - Investigational Site Number 1520005, Santiago
  - Investigational Site Number 1520012, Santiago
  - Investigational Site Number 1520013, Santiago
  - Investigational Site Number 1520002, Temuco
  - Investigational Site Number 1520001, Viña del Mar
  - Investigational Site Number 1520010, Viña del Mar
- Czechia (14):
  - Investigational Site Number 2030001, Brno
  - Investigational Site Number 2030003, Brno
  - Investigational Site Number 2030004, Brno
  - Investigational Site Number 2030014, Kolín
  - Investigational Site Number 2030010, Kroměříž
  - Investigational Site Number 2030005, Liberec
  - Investigational Site Number 2030013, Městec Králové
  - Investigational Site Number 2030018, Prague
  - Investigational Site Number 2030002, Prague
  - Investigational Site Number 2030017, Prague
  - Investigational Site Number 2030007, Praha 5 - Motol
  - Investigational Site Number 2030015, Pribram I
  - Investigational Site Number 2030011, Přerov
  - Investigational Site Number 2030006, Slaný
- Denmark (5):
  - Investigational Site Number 2080004, Aalborg
  - Investigational Site Number 2080003, Aarhus N
  - Investigational Site Number 2080002, Glostrup Municipality
  - Investigational Site Number 2080001, Herlev
  - Investigational Site Number 2080005, København NV
- Finland (5):
  - Investigational Site Number 2460004, Espoo
  - Investigational Site Number 2460001, Helsinki
  - Investigational Site Number 2460002, Jyväskylä
  - Investigational Site Number 2460003, Oulu
  - Investigational Site Number 2460005, Seinäjoki
- France (11):
  - Investigational Site Number 2500009, Chambray-lès-Tours
  - Investigational Site Number 2500008, La Tronche
  - Investigational Site Number 2500004, Le Chesnay
  - Investigational Site Number 2500002, Le Coudray
  - Investigational Site Number 2500001, Lille
  - Investigational Site Number 2500007, Nantes
  - Investigational Site Number 2500012, Nice
  - Investigational Site Number 2500006, Paris
  - Investigational Site Number 2500003, Paris
  - Investigational Site Number 2500005, Toulouse
  - Investigational Site Number 2500013, Vandœuvre-lès-Nancy
- Germany (29):
  - Investigational Site Number 2760020, Bad Nauheim
  - Investigational Site Number 2760016, Bad Oeynhausen
  - Investigational Site Number 2760013, Berlin
  - Investigational Site Number 2760019, Berlin
  - Investigational Site Number 2760001, Berlin
  - Investigational Site Number 2760002, Berlin
  - Investigational Site Number 2760025, Bielefeld
  - Investigational Site Number 2760005, Bonn
  - Investigational Site Number 2760021, Bremen
  - Investigational Site Number 2760035, Coburg
  - Investigational Site Number 2760027, Cologne
  - Investigational Site Number 2760032, Dortmund
  - Investigational Site Number 2760006, Dortmund
  - Investigational Site Number 2760029, Erfurt
  - Investigational Site Number 2760018, Essen
  - Investigational Site Number 2760033, Frankfurt am Main
  - Investigational Site Number 2760009, Greifswald
  - Investigational Site Number 2760022, Heidelberg
  - Investigational Site Number 2760031, Heidelberg
  - Investigational Site Number 2760034, Lahr
  - Investigational Site Number 2760030, Langen
  - Investigational Site Number 2760014, Leverkusen
  - Investigational Site Number 2760036, Limburg
  - Investigational Site Number 2760012, Ludwigshafen
  - Investigational Site Number 2760028, Merseburg
  - Investigational Site Number 2760011, Rotenburg an der Fulda
  - Investigational Site Number 2760015, Rüsselsheim am Main
  - Investigational Site Number 2760007, Witten
  - Investigational Site Number 2760026, Würzburg
- Greece (10):
  - Investigational Site Number 3000012, Athens
  - Investigational Site Number 3000004, Athens
  - Investigational Site Number 3000002, Chalcis
  - Investigational Site Number 3000009, Elefsina
  - Investigational Site Number 3000003, Haidari
  - Investigational Site Number 3000005, Heraklion
  - Investigational Site Number 3000007, Ioannina
  - Investigational Site Number 3000006, Larissa
  - Investigational Site Number 3000001, N. Ionia
  - Investigational Site Number 3000008, Thessaloniki
- Hungary (19):
  - Investigational Site Number 3480018, Berettyóújfalu
  - Investigational Site Number 3480012, Budapest
  - Investigational Site Number 3480016, Budapest
  - Investigational Site Number 3480010, Budapest
  - Investigational Site Number 3480019, Budapest
  - Investigational Site Number 3480001, Budapest
  - Investigational Site Number 3480015, Budapest
  - Investigational Site Number 3480011, Budapest
  - Investigational Site Number 3480014, Budapest
  - Investigational Site Number 3480005, Budapest
  - Investigational Site Number 3480007, Debrecen
  - Investigational Site Number 3480002, Dombóvár
  - Investigational Site Number 3480017, Gyula
  - Investigational Site Number 3480008, Hódmezövásárhely
  - Investigational Site Number 3480020, Kistarcsa
  - Investigational Site Number 3480009, Komárom
  - Investigational Site Number 3480013, Pécs
  - Investigational Site Number 3480003, Székesfehérvár
  - Investigational Site Number 3480006, Zalaegerszeg
- Israel (12):
  - Investigational Site Number 3760013, Ashkelon
  - Investigational Site Number 3760004, Hadera
  - Investigational Site Number 3760005, Haifa
  - Investigational Site Number 3760006, Jerusalem
  - Investigational Site Number 3760003, Jerusalem
  - Investigational Site Number 3760008, Jerusalem
  - Investigational Site Number 3760010, Nahariya
  - Investigational Site Number 3760002, Petah Tikva
  - Investigational Site Number 3760011, Rehovot
  - Investigational Site Number 3760009, Safed
  - Investigational Site Number 3760001, Tel Aviv
  - Investigational Site Number 3760012, Tiberias
- Italy (21):
  - Investigational Site Number 3800006, Arzignano (Vi)
  - Investigational Site Number 3800011, Brescia
  - Investigational Site Number 3800017, Brescia
  - Investigational Site Number 3800005, Cortona
  - Investigational Site Number 3800009, Ferrara
  - Investigational Site Number 3800020, Gallipoli
  - Investigational Site Number 3800003, Legnago
  - Investigational Site Number 3800023, Milan
  - Investigational Site Number 3800002, Milan
  - Investigational Site Number 3800012, Milan
  - Investigational Site Number 3800008, Milan
  - Investigational Site Number 3800013, Monza
  - Investigational Site Number 3800022, Napoli
  - Investigational Site Number 3800018, Pavia
  - Investigational Site Number 3800004, Perugia
  - Investigational Site Number 3800016, Pozzilli
  - Investigational Site Number 3800014, Rimini
  - Investigational Site Number 3800010, Roma
  - Investigational Site Number 3800021, Roma
  - Investigational Site Number 3800019, Scorrano
  - Investigational Site Number 3800007, Udine
- Latvia (4):
  - Investigational Site Number 4280004, Daugavpils
  - Investigational Site Number 4280002, Liepāja
  - Investigational Site Number 4280001, Riga
  - Investigational Site Number 4280003, Riga
- Lithuania (6):
  - Investigational Site Number 4400002, Kaunas
  - Investigational Site Number 4400005, Kaunas
  - Investigational Site Number 4400004, Klaipėda
  - Investigational Site Number 4400006, Šiauliai
  - Investigational Site Number 4400001, Vilnius
  - Investigational Site Number 4400003, Vilnius
- Netherlands (8):
  - Investigational Site Number 5280004, 's-Hertogenbosch
  - Investigational Site Number 5280003, Amsterdam
  - Investigational Site Number 5280001, Breda
  - Investigational Site Number 5280007, Delft
  - Investigational Site Number 5280002, Doetinchem
  - Investigational Site Number 5280006, Rotterdam
  - Investigational Site Number 5280008, Sneek
  - Investigational Site Number 5280005, Veldhoven
- New Zealand (6):
  - Investigational Site Number 5540007, Auckland
  - Investigational Site Number 5540006, Christchurch
  - Investigational Site Number 5540002, Hamilton
  - Investigational Site Number 5540004, Lower Hutt
  - Investigational Site Number 5540005, New Plymouth
  - Investigational Site Number 5540003, Rotorua
- Poland (19):
  - Investigational Site Number 6160007, Bialystok
  - Investigational Site Number 6160017, Gdansk
  - Investigational Site Number 6160002, Grodzisk Mazowiecki
  - Investigational Site Number 6160014, Katowice
  - Investigational Site Number 6160021, Krakow
  - Investigational Site Number 6160001, Krakow
  - Investigational Site Number 6160003, Krakow
  - Investigational Site Number 6160012, Krakow
  - Investigational Site Number 6160016, Lubin
  - Investigational Site Number 6160005, Miechów
  - Investigational Site Number 6160022, Poznan
  - Investigational Site Number 6160006, Torun
  - Investigational Site Number 6160013, Warsaw
  - Investigational Site Number 6160004, Warsaw
  - Investigational Site Number 6160020, Warsaw
  - Investigational Site Number 6160024, Warsaw
  - Investigational Site Number 6160008, Warsaw
  - Investigational Site Number 6160015, Zamość
  - Investigational Site Number 6160011, Łęczna
- Portugal (10):
  - Investigational Site Number 6200012, Braga
  - Investigational Site Number 6200001, Coimbra
  - Investigational Site Number 6200011, Guilhufe - Penafiel
  - Investigational Site Number 6200004, Guimarães
  - Investigational Site Number 6200006, Lisbon
  - Investigational Site Number 6200002, Lisbon
  - Investigational Site Number 6200008, Porto
  - Investigational Site Number 6200007, Vila Franca de Xira
  - Investigational Site Number 6200003, Vila Nova Gaia
  - Investigational Site Number 6200005, Vila Real
- Romania (18):
  - Investigational Site Number 6420014, Arad
  - Investigational Site Number 6420006, Baia Mare
  - Investigational Site Number 6420015, Brăila
  - Investigational Site Number 6420013, Bucharest
  - Investigational Site Number 6420019, Bucharest
  - Investigational Site Number 6420011, Bucharest
  - Investigational Site Number 6420008, Bucharest
  - Investigational Site Number 6420007, Bucharest
  - Investigational Site Number 6420002, Cluj-Napoca
  - Investigational Site Number 6420003, Cluj-Napoca
  - Investigational Site Number 6420016, Craiova
  - Investigational Site Number 6420005, Oradea
  - Investigational Site Number 6420004, Oradea
  - Investigational Site Number 6420018, Satu Mare
  - Investigational Site Number 6420001, Târgu Mureş
  - Investigational Site Number 6420012, Tg-Mures
  - Investigational Site Number 6420009, Timișoara
  - Investigational Site Number 6420010, Timișoara
- Russia (20):
  - Investigational Site Number 6430026, Ivanovo
  - Investigational Site Number 6430023, Kazan'
  - Investigational Site Number 6430002, Kemerovo
  - Investigational Site Number 6430006, Kemerovo
  - Investigational Site Number 6430005, Moscow
  - Investigational Site Number 6430004, Moscow
  - Investigational Site Number 6430022, Moscow
  - Investigational Site Number 6430024, Moscow
  - Investigational Site Number 6430001, Moscow
  - Investigational Site Number 6430003, Moscow
  - Investigational Site Number 6430010, Moscow
  - Investigational Site Number 6430018, Nizhny Novgorod
  - Investigational Site Number 6430013, Rostov-on-Don
  - Investigational Site Number 6430025, Saint Petersburg
  - Investigational Site Number 6430007, Saint Petersburg
  - Investigational Site Number 6430012, Saint Petersburg
  - Investigational Site Number 6430011, Saint Petersburg
  - Investigational Site Number 6430009, Saint Petersburg
  - Investigational Site Number 6430017, Sochi
  - Investigational Site Number 6430016, Tomsk
- Slovakia (8):
  - Investigational Site Number 7030001, Bratislava
  - Investigational Site Number 7030004, Bratislava
  - Investigational Site Number 7030003, Bratislava 3 - Kramare
  - Investigational Site Number 7030010, Brezno
  - Investigational Site Number 7030009, Dolný Kubín
  - Investigational Site Number 7030002, Košice
  - Investigational Site Number 7030011, Nitra
  - Investigational Site Number 7030008, Trnava
- South Korea (10):
  - Investigational Site Number 4100008, Bucheon-si
  - Investigational Site Number 4100010, Busan
  - Investigational Site Number 4100004, Daegu
  - Investigational Site Number 4100001, Hwaseong-si
  - Investigational Site Number 4100003, Incheon
  - Investigational Site Number 4100005, Seongnam-si
  - Investigational Site Number 4100002, Seoul
  - Investigational Site Number 4100007, Seoul
  - Investigational Site Number 4100011, Seoul
  - Investigational Site Number 4100009, Seoul
- Spain (21):
  - Investigational Site Number 7240006, A Coruña
  - Investigational Site Number 7240016, Alicante
  - Investigational Site Number 7240015, Badalona
  - Investigational Site Number 7240020, L'Hospitalet de Llobregat
  - Investigational Site Number 7240005, Las Palmas de Gran Canaria
  - Investigational Site Number 7240021, Madrid
  - Investigational Site Number 7240008, Madrid
  - Investigational Site Number 7240022, Manises
  - Investigational Site Number 7240004, Málaga
  - Investigational Site Number 7240007, Murcia
  - Investigational Site Number 7240014, Olot
  - Investigational Site Number 7240009, San Sebastián de los Reyes
  - Investigational Site Number 7240003, Sanlúcar de Barrameda
  - Investigational Site Number 7240001, Seville
  - Investigational Site Number 7240019, Seville
  - Investigational Site Number 7240018, Úbeda
  - Investigational Site Number 7240012, Valencia
  - Investigational Site Number 7240011, Valencia
  - Investigational Site Number 7240010, Valencia
  - Investigational Site Number 7240002, Villamartín
  - Investigational Site Number 7240013, Zaragoza
- Sweden (6):
  - Investigational Site Number 7520004, Jönköping
  - Investigational Site Number 7520002, Malmo
  - Investigational Site Number 7520006, Skellefteå
  - Investigational Site Number 7520007, Stockholm
  - Investigational Site Number 7520008, Stockholm
  - Investigational Site Number 7520001, Stockholm
- Switzerland (2):
  - Investigational Site Number 7560001, Basel
  - Investigational Site Number 7560003, Lugano
- Turkey (Türkiye) (10):
  - Investigational Site Number 7920008, Antalya
  - Investigational Site Number 7920006, Çorum
  - Investigational Site Number 7920005, Eskişehir
  - Investigational Site Number 7920002, Haseki/ Istanbul
  - Investigational Site Number 7920011, Istanbul
  - Investigational Site Number 7920012, Izmir
  - Investigational Site Number 7920003, Kocaeli
  - Investigational Site Number 7920004, Mersin
  - Investigational Site Number 7920001, Sivas
  - Investigational Site Number 7920010, Trabzon
- United Kingdom (10):
  - Investigational Site Number 8260005, Bournemouth
  - Investigational Site Number 8260010, Bristol
  - Investigational Site Number 8260008, Chelmsford
  - Investigational Site Number 8260009, Hull
  - Investigational Site Number 8260002, Newcastle
  - Investigational Site Number 8260001, Oldham
  - Investigational Site Number 8260003, Swansea
  - Investigational Site Number 8260006, Swindon
  - Investigational Site Number 8260004, Torquay
  - Investigational Site Number 8260007, York

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants.

REFERENCES:
- [Derived] Bhatt AS, Bhatt DL, Steg PG, Szarek M, Cannon CP, Leiter LA, McGuire DK, Lewis JB, Riddle MC, Voors AA, Metra M, Lund LH, Testani JM, Wilcox CS, Davies M, Pitt B, Kosiborod MN. Effects of Sotagliflozin on Health Status in Patients With Worsening Heart Failure: Results From SOLOIST-WHF. J Am Coll Cardiol. 2024 Sep 17;84(12):1078-1088. doi: 10.1016/j.jacc.2024.06.036. PMID 39260929
- [Derived] Weintraub WS, Kolm P, Dolman S, Alva M, Bhatt DL, Zhang Z. Cost-Effectiveness of Sotagliflozin in SOLOIST-WHF. JACC Heart Fail. 2024 Sep;12(9):1600-1610. doi: 10.1016/j.jchf.2024.04.018. Epub 2024 Jun 12. PMID 38878007
- [Derived] Kim J, Wang S, Sikirica S, Shafrin J. Cost-effectiveness of sotagliflozin for the treatment of patients with diabetes and recent worsening heart failure. J Comp Eff Res. 2024 Jun;13(6):e230190. doi: 10.57264/cer-2023-0190. Epub 2024 May 21. PMID 38771012
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Szarek M, Bhatt DL, Steg PG, Cannon CP, Leiter LA, McGuire DK, Lewis JB, Riddle MC, Voors AA, Metra M, Lund LH, Komajda M, Testani JM, Wilcox CS, Ponikowski P, Lopes RD, Banks P, Tesfaye E, Ezekowitz JA, Verma S, Pitt B; SOLOIST-WHF committees and investigators. Effect of Sotagliflozin on Total Hospitalizations in Patients With Type 2 Diabetes and Worsening Heart Failure : A Randomized Trial. Ann Intern Med. 2021 Aug;174(8):1065-1072. doi: 10.7326/M21-0651. Epub 2021 Jun 22. PMID 34152828
- [Derived] Bhatt DL, Szarek M, Steg PG, Cannon CP, Leiter LA, McGuire DK, Lewis JB, Riddle MC, Voors AA, Metra M, Lund LH, Komajda M, Testani JM, Wilcox CS, Ponikowski P, Lopes RD, Verma S, Lapuerta P, Pitt B; SOLOIST-WHF Trial Investigators. Sotagliflozin in Patients with Diabetes and Recent Worsening Heart Failure. N Engl J Med. 2021 Jan 14;384(2):117-128. doi: 10.1056/NEJMoa2030183. Epub 2020 Nov 16. PMID 33200892

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 306 investigative sites in North America, Latin America, Western Europe, Eastern Europe, and the Rest of the World from 15 June 2018 to 05 June 2020.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes post Worsening Heart Failure were enrolled equally in 1 of 2 treatment groups, sotagliflozin or placebo.
Period: Overall Study
Arm/Group | Sotagliflozin | Placebo
Started | 608 | 614
Randomized and Treated | 605 | 611
Completed | 0 | 0
Not Completed | 608 | 614
Not completed — Death | 65 | 73
Not completed — Withdrawal by Subject | 18 | 23
Not completed — Site Terminated by Sponsor | 39 | 35
Not completed — Study Terminated by Sponsor | 483 | 477
Not completed — Reason not Specified | 3 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sotagliflozin | Placebo | Total
Number analyzed (Participants) | 608 | 614 | 1222
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (9.5) | 69.3 (8.8) | 68.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 214 | 412
  Male | 410 | 400 | 810
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 163 | 157 | 320
  Not Hispanic or Latino | 438 | 455 | 893
  Unknown or Not Reported | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 25 | 25 | 50
  White | 567 | 572 | 1139
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Total Occurrences of Cardiovascular (CV) Death, Hospitalizations for Heart Failure (HHF) and Urgent Visits for Heart Failure (HF)
Description: Combined endpoint of the total number of occurrences (first and potentially subsequent) of CV death, HHF, and urgent HF visits after randomization. Events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 21.9 months
Population: ITT population includes all randomized participants.
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 608 | 614
events per 100-person years | 51 | 76.3
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; The estimates of the hazard ratio (HR) and corresponding 2-sided 95% confidence interval (CI) was to be provided by a marginal Cox proportional hazard model stratified by region and ejection fraction, with non-cardiovascular (non-CV) death treated as a competing event; Test type: Superiority; p < 0.001, Cox proportional hazards model; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.52 to 0.85]

2. Secondary Outcome: Total Number of Occurrences of HHF and Urgent HF Visits
Description: Combined endpoint of the total occurrences (first and potentially subsequent) of HHF and urgent HF visits after randomization. Events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 21.9 months
Population: ITT population includes all randomized participants.
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 608 | 614
events per 100-person years | 40.4 | 63.9
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; The estimates of the HR and corresponding 2-sided 95% CI was to be provided by a marginal Cox proportional hazard model stratified by region and ejection fraction, with non-CV death treated as a competing event; Test type: Superiority; p < 0.001, Cox proportional hazards model; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.49 to 0.83]

3. Secondary Outcome: Total Number of Deaths From Cardiovascular Causes
Description: Number of events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 21.9 months
Population: ITT population includes all randomized participants.
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 608 | 614
events per 100-person years | 10.6 | 12.5
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.36, Cox proportional hazards model; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.58 to 1.22]

4. Secondary Outcome: Total Number of Occurrences of CV Death, HHF, Non-fatal Myocardial Infarction and Non-fatal Stroke
Description: Combined endpoint of the total number of occurrences (first and potentially subsequent) of CV death, HHF, non-fatal stroke, and non-fatal myocardial infarction after randomisation. Events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 21.9 months
Population: ITT population includes all randomized participants.
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 608 | 614
events per 100-person years | 51.4 | 71.0
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.56 to 0.92]

5. Secondary Outcome: Total Number of Occurrences of HHF, Urgent HF Visit, CV Death, and HF While Hospitalized
Description: Combined endpoint of the total number of occurrences (first and potentially subsequent) after randomisation of HHF, urgent HF visits, CV Death and HF while hospitalised. Events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 21.9 months
Population: ITT population includes all randomized participants.
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 608 | 614
events per 100-person years | 54.7 | 80.6
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.54 to 0.86]

6. Secondary Outcome: Total Number of Deaths From Any Cause
Description: as for outcome 3
Time Frame: Up to 21.9 months
Population: ITT population includes all randomized participants.
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 608 | 614
events per 100-person years | 13.5 | 16.3
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; The estimates of the HR and corresponding 2-sided 95% CI was to be provided by a marginal Cox proportional hazard model stratified by region and ejection fraction; Test type: Superiority; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.59 to 1.14]

7. Secondary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12) Scores at Month 4
Description: KCCQ-12 is a 12 question questionnaire, participants completed questionnaire about how heart failure affected their life over the past 2 weeks. The scale has 4 domains: symptom frequency, physical limitation, social limitations and quality of life for a total possible transformed score of 0 to 100 where 100 denotes the highest health status. A positive change from baseline indicates improvement. An analysis of covariance (ANCOVA) model was used for analysis.
Time Frame: Baseline to Month 4
Population: ITT population includes all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 608 | 614
score on a scale | 17.7 (0.41) | 13.6 (0.41)
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; The change from baseline to Month 4 was analyzed using an ANCOVA model with treatment groups as factor and baseline KCCQ-12 score and randomization stratification factors as covariates; Test type: Superiority; Hazard Ratio (HR) = 4.1, 95% CI 2-sided [1.3 to 7]

8. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR is a test for renal function. A blood sample was collected and was sent to a central laboratory. eGFR was calculated by the Modification of Diet in Renal Disease (MDRD) equation reported as milliliters/minute/1.73 meter squared (mL/min/1.73 m^2). A mixed model for repeated measures (MMRM) was used for analysis.
Time Frame: Baseline up to 21.9 months
Population: ITT population includes all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73 m^2
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 608 | 614
mL/min/1.73 m^2 | -0.34 (1.33) | -0.18 (1.33)
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; Rate of decline in eGFR observed over time was analyzed by MMRM with absolute change in eGFR from baseline as the outcome, a random effect for intercept, and fixed effects for treatment, baseline value, and time; Test type: Superiority; Difference in Least Squares Means = -0.16, 95% CI 2-sided [-1.3 to 0.98]

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 10 days after the last dose of study drug (Up to 21.9 months)
Description: Number of Deaths (All causes) is based on all randomized participants (n=608,614). Adverse Events are based on the Safety population that included all randomized participants who received at least one dose of study drug (n=605,611).
Arm/Group | Sotagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 65/608 | 76/614
Serious Adverse Events (participants affected / at risk) | 235/605 | 251/611
Other Adverse Events (participants affected / at risk) | 101/605 | 90/611
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sotagliflozin (N=605) | Placebo (N=611)
Aortic rupture (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 6 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 5
Peripheral artery occlusion (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 2 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1
Aortic valve replacement (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 0
Cardiac rehabilitation therapy (Surgical and medical procedures) | 1 | 1
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1
Therapeutic procedure (Surgical and medical procedures) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Asthenia (General disorders) | 0 | 1
Cardiac death (General disorders) | 0 | 1
Chest pain (General disorders) | 3 | 0
Death (General disorders) | 2 | 4
Fatigue (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Nodule (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 3
Sudden cardiac death (General disorders) | 7 | 9
Sudden death (General disorders) | 2 | 2
Vascular stent thrombosis (General disorders) | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 3
Drug abuse (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Biopsy prostate (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Catheterisation cardiac (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Liver function test increased (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Transplant evaluation (Investigations) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 2 | 2
Acute myocardial infarction (Cardiac disorders) | 4 | 3
Angina pectoris (Cardiac disorders) | 4 | 3
Angina unstable (Cardiac disorders) | 8 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 8 | 8
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 80 | 121
Cardiac failure acute (Cardiac disorders) | 12 | 11
Cardiac failure chronic (Cardiac disorders) | 1 | 8
Cardiac failure congestive (Cardiac disorders) | 11 | 16
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 2 | 2
Chronic left ventricular failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 6 | 9
Myocardial ischaemia (Cardiac disorders) | 2 | 1
Pericardial effusion (Cardiac disorders) | 0 | 2
Pericarditis (Cardiac disorders) | 2 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Sinoatrial block (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 4 | 4
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 7
Brain oedema (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 5 | 3
Cognitive disorder (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 9 | 9
Loss of consciousness (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Postresuscitation encephalopathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 0 | 1
Spinal cord ischaemia (Nervous system disorders) | 1 | 0
Spinal cord ischaemia Syncope (Nervous system disorders) | 2 | 12
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Eye haemorrhage (Eye disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Splenic artery aneurysm (Gastrointestinal disorders) | 0 | 1
Ulcerative gastritis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 11 | 16
Calculus urinary (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 3 | 6
Haematuria (Renal and urinary disorders) | 1 | 1
Nephritis (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 6
Renal impairment (Renal and urinary disorders) | 0 | 3
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 2
Device malfunction (Product Issues) | 1 | 1
Lead dislodgement (Product Issues) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2
Bronchitis viral (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 4 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Infective thrombosis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pharyngeal abscess (Infections and infestations) | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 19 | 26
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 0 | 4
Septic shock (Infections and infestations) | 2 | 4
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 6
Urosepsis (Infections and infestations) | 3 | 1
Viral infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sotagliflozin (N=605) | Placebo (N=611)
Hypotension (Vascular disorders) | 33 | 27
Cardiac failure (Cardiac disorders) | 41 | 57
Diarrhoea (Gastrointestinal disorders) | 36 | 18

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of participants analyzed or technical problems leading to unreliable data.

The study was terminated prematurely due to business decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT03521934/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03521934/SAP_001.pdf